CLINICAL TRIAL: NCT02598011
Title: The Toca 7 Study: A Phase 1b Study of the Safety of Toca 511, a Retroviral Replicating Vector, Combined With Toca FC in Subjects With Newly Diagnosed High Grade Glioma Receiving Standard of Care
Brief Title: A Study of the Safety of Toca 511, a Retroviral Replicating Vector, Combined With Toca FC in Subjects With Newly Diagnosed High Grade Glioma Receiving Standard of Care
Acronym: Toca7
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Tocagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tg 511-15-03
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2015-12

CONDITIONS: Newly Diagnosed High Grade Glioma (HGG)
MeSH Terms: interventions — vocimagene amiretrorepvec; Flucytosine

ARMS (2):
- Toca 511/Toca FC at 170 mg/kg/day (Experimental): Toca 511: 4 mL administered by intracranial parenchymal injection into the walls of the resection cavity following tumor resection or, for those subjects who are not candidates for resection, via stereotactic injection into their tumor using a standard Nashold-type side cutting biopsy needle.
  Toca FC: Approximately 4 to 6 weeks after tumor resection, subjects will begin temozolomide concurrent with radiation therapy. During concurrent chemoradiation at the start of the second and sixth week of concurrent chemoradiation and every 28 days thereafter, a 7-day course of oral Toca FC will be dosed at 170 mg/kg/day
  Interventions: Biological: Toca 511; Drug: Toca FC
- Toca 511/Toca FC at 220 mg/kg/day (Experimental): Toca 511: 4 mL administered by intracranial parenchymal injection into the walls of the resection cavity following tumor resection or, for those subjects who are not candidates for resection, via stereotactic injection into their tumor using a standard Nashold-type side cutting biopsy needle.
  Toca FC: Approximately 4 to 6 weeks after tumor resection, subjects will begin temozolomide concurrent with radiation therapy. During concurrent chemoradiation at the start of the second and sixth week of concurrent chemoradiation and every 28 days thereafter, a 7-day course of oral Toca FC will be dosed at 220 mg/kg/day
  Interventions: Biological: Toca 511; Drug: Toca FC

INTERVENTIONS:
Biological: Toca 511 — Toca 511 consists of a purified retroviral replicating vector encoding a modified yeast cytosine deaminase (CD) gene. The CD gene converts the antifungal 5-flurocytosine (5FC) to the anticancer drug 5-FU in cells that have been infected by the Toca 511 vector
  Other Names: vocimagene amiretrorepvec; RRV; retroviral replicating viral
Drug: Toca FC — Toca FC is an extended-release formulation of flucytosine. Toca FC is supplied as 500 mg white, oblong tablets with "TOCA FC" embossed on one side and "500" embossed on the other side
  Other Names: Flucytosine; 5-FC; 5-Fluorocytosine

SUMMARY:
This is a multi-center, open label trial of combination therapy with Toca 511 and ascending doses of Toca FC added to the SOC for newly diagnosed HGG.

DETAILED DESCRIPTION:
This is a multi-center, open label trial of combination therapy with Toca 511 and ascending doses of Toca FC added to the SOC for newly diagnosed HGG.

Enrolled subjects with presumed newly diagnosed HGG will undergo planned resection of tumor.

Subjects with HGG will receive Toca 511, administered by intracranial parenchymal injection into the walls of the resection cavity.

This study will establish the recommended Phase 2 dose of Toca FC to be used in combination with standard of care chemoradiation and temozolomide in subjects with newly diagnosed HGG.

Subjects will begin chemoradiation treatment approximately 4 to 6 weeks after surgery. Oral Toca FC (7-day courses) will be administered concurrent with the start of the second and sixth weeks of chemoradiation during the concurrent treatment period, and concurrent with the start of temozolomide during the maintenance treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given written informed consent
2. Subject is at least 18 years old
3. Subjects must have presumed newly diagnosed high grade glioma prior to tissue diagnosis or definitive initial surgical resection
4. Based on the pre-operative evaluation by neurosurgeon, the subject is a candidate for planned resection of enhancing region of tumor OR for those subjects who are not candidates for resection, based on the pre-operative evaluation by neurosurgeon, the subject has a presumed newly diagnosed high grade glioma accessible by a technically feasible stereotactic trajectory
5. Laboratory values adequate for subject to undergo surgery, including:

   * Platelet count ≥ 100,000/mm3
   * Hgb ≥ 10 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,500/mm3
   * Normal PT/PTT (subnormal PT/PTT acceptable)
   * Adequate liver function, including total bilirubin ≤ 1.5 x ULN (unless known Gilbert's syndrome); ALT ≤ 2.5 x ULN
6. The subject has a KPS ≥ 70
7. Women of childbearing potential (≥12 months of non-therapy-induced amenorrhea or surgically sterile) must have had a negative serum pregnancy test within the past 21 days and must use a birth control method in addition to barrier methods (condoms)
8. Subject or subject's partner is willing to use condoms for 12 months after receiving Toca 511 or until there is no evidence of the virus in his/her blood, whichever is longer
9. Subject has an absolute lymphocyte count (ALC) ≥ 500/mm3
10. Estimated glomerular filtration rate of at least 50 mL/min by the Cockcroft Gault formula

Exclusion Criteria:

1. History of other malignancy, unless the subject has been disease free for at least 5 years. Adequately treated basal cell carcinoma or squamous cell skin cancer is acceptable regardless of time, as well as localized prostate carcinoma or cervical carcinoma in situ after curative treatment
2. A contrast enhancing brain tumor that is any of the following:

   * Multi focal (defined as 2 separate areas of contrast enhancement measuring at least 1 cm in 2 planes that are not contiguous on either fluid attenuated inversion recovery (FLAIR) or T2 sequences);
   * Associated with either diffuse subependymal or leptomeningeal dissemination; or > 5 cm in any dimension
   * Location in the brainstem, cerebellum or spinal cord

   Expansion Cohort:

   OR For those subjects who are not candidates for resection, injection of the tumor requires violation of the ventricular system
3. The subject has or had any active infection requiring antibiotic, antifungal or antiviral therapy within the past 4 weeks
4. The subject has any bleeding diathesis, or must take anticoagulants, or antiplatelet agents, including nonsteroidal anti-inflammatory drugs (NSAIDs), at the time of the scheduled surgery that cannot be stopped for surgery
5. The subject received any investigational treatment for any reason within the past 30 days. Investigational agents used to improve surgical resection or craniotomy wound healing or recovery are allowed.
6. The subject intends to undergo treatment with the Gliadel® wafer at the time of this surgery
7. Prior intracranial gamma knife, stereotactic radiosurgery, or other focal high-dose radiotherapy is not allowed
8. Severe pulmonary, cardiac or other systemic disease, specifically:

   * New York Heart Association > Grade 2 congestive heart failure within 6 months prior to study entry, unless asymptomatic and well controlled with medication (see Appendix G)
   * Uncontrolled or significant cardiovascular disease, clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or Torsades des pointes), clinically significant pulmonary disease (such as ≥ Grade 2 dyspnea, according to CTCAE 4.03)
   * Subjects who have any other disease, either metabolic or psychological, which as per Investigator assessment may affect the subject's compliance or place the subject at higher risk of potential treatment complications
9. The subject is breast feeding
10. The subject is HIV positive
11. The subject has a history of allergy or intolerance to flucytosine
12. The subject has a gastrointestinal disease that would prevent him or her from being able to swallow Toca FC tablets or absorb flucytosine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities | 12 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.felt to be related to Toca 511 or the Toca 511/5-FC combination